CLINICAL TRIAL: NCT05820698
Title: A Feasibility Pilot Study Examining the Effect of a Mediterranean Style Diet and Time-restricted Eating on Individuals With Mild-moderate Psoriasis
Brief Title: The Mediterranean Diet and Time-Restricted Eating Dietary Interventions for Psoriasis Study
Acronym: METRED-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Psoriasis Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR/DP-22/23-34784
Record Dates: First submitted 2023-03-16; First posted 2023-04-20 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis Vulgaris
Keywords: Diet; Inflammation; Mediterranean diet; Time-restricted eating; Nutrition
MeSH Terms: conditions — Inflammation; Intermittent Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Given the nature of dietary interventions, blinding will not always be possible, and this study will be conducted in an unblinded manner. Only the Consultant Dermatologist (Outcome Assessor) undertaking the psoriasis severity examinations will be blinded to the allocated diet interventions of the participants. All statistical data analysis will be carried out blinded using data codes to ensure that the intervention allocation is concealed from the researcher carrying out the statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The Mediterranean style diet (Experimental): Participants in the Mediterranean style diet arm (n = 12) will receive dietary advice to follow a Mediterranean style diet by the Research Nutritionist.
  Interventions: Other: The Mediterranean style diet
- The Mediterranean style diet with time-restricted eating (Experimental): Participants in the Mediterranean style diet with time-restricted eating arm (n = 12) will receive dietary advice to follow a Mediterranean style diet combined with time-restricted eating by the Research Nutritionist.
  Interventions: Other: The Mediterranean style diet; Other: Time-restricted eating
- The UK diet with time-restricted eating (Active Comparator): Participants in the UK diet with time-restricted eating arm (n = 12) will receive dietary advice to follow a UK diet combined with time-restricted eating by the Research Nutritionist.
  Interventions: Other: The UK diet; Other: Time-restricted eating

INTERVENTIONS:
Other: The Mediterranean style diet — Participants in the Mediterranean style diet group will be provided with recommendations to include a minimum of 5 servings of fruits and vegetables (combined) per day, 2 servings of whole grains per meal per day, at least two servings of extra virgin olive oil per day, a maximum two servings of dairy products per day (excluding milk in coffee/tea), a minimum of 3 servings of fish per week (of which two should be oily fish), less than 2 servings of red meat or processed meat per week. Confectionary and sugar sweetened beverages should be limited to less than 2 servings per week.
  Participants randomised to the Mediterranean style intervention will be provided with support documents including a dietary guideline booklet, recipes, meal plans, shopping and product swap lists, as well as eating-out and budget-eating advice sheets. Food deliveries containing key food items of the diet intervention will be scheduled for week 1, week 4, and week 8 of the study.
  Arms: The Mediterranean style diet; The Mediterranean style diet with time-restricted eating
Other: The UK diet — Participants in the UK diet with time-restricted eating group will be provided with recommendations of a nutritionally balanced diet, corresponding to the average intakes of the UK population. Participants will be advised to consume no more than 4 portions of fruits and vegetables combined per day, to have at least two servings of dairy per day, to limit the consumption of white fish to less than 1 serving per week, with ≤1 serving of oily fish per month. Nuts and seeds consumption should also be limited to ≤1 serving per week and at least 3 servings of white and red meat should be consumed per week.
  Participants randomised to the UK diet will be provided with support documents including a dietary guideline booklet, recipes, and meal plans. A £30 reimbursement will be provided to participants for their grocery shopping on week 1, week 4, and week 8 of the study.
  Arms: The UK diet with time-restricted eating
Other: Time-restricted eating — Participants randomised to the time-restricted eating interventions will be advised to limit food intake to a 10-hour eating window and to abstain from food intake for a 14-hour fasting window. Hydration is to be maintained during the fasting window with water and/or plain teas/coffees
  Arms: The Mediterranean style diet with time-restricted eating; The UK diet with time-restricted eating

SUMMARY:
The METRED-P study will test the feasibility of implementing a Mediterranean style diet and/or time-restricted eating as dietary patterns in individuals with psoriasis. This study will address the following research questions:

1. Are participants' able to adhere to the allocated dietary intervention?
2. What is the participants' acceptability of the allocated dietary intervention?
3. What is the practicality (from a clinician's stand point) of delivering the dietary interventions?
4. When adhering to the allocated intervention, are there changes in psoriasis severity?
5. When adhering to the allocated intervention, are there changes in measures of body composition?
6. When adhering to the allocated intervention, are there changes in fasting blood measures?

Participants will attend an initial clinic visit for a fasting blood sample, psoriasis examination, body composition measurements, and will complete short multiple-choice questionnaires on the severity of their psoriasis. A Research Nutritionist will deliver the diet interventions as diet consultation sessions. These sessions are reoccurring throughout the study as virtual consultation booster sessions, which are supplemented with wellbeing check-in calls. Participants will complete short questionnaires on the severity of their psoriasis and will record their dietary intake for 4 days, before the start of the study, and on week 1, week 6, and week 12 of the study. The allocated diet should be adhered to for 12 weeks until the end of the study, where participants will return and attend a final clinic visit to repeat the measures obtained during the initial clinic visit.

Researchers will compare the feasibility of implementing a Mediterranean style diet and a Mediterranean style diet with time-restricted eating, with a UK diet with time-restricted eating.

DETAILED DESCRIPTION:
The METRED-P study is a 12-week dietary intervention in individuals with mild-moderate psoriasis. Participants will be randomly allocated to one of three groups: a Mediterranean style diet only, a Mediterranean style diet with time-restricted eating or a UK diet with time-restricted eating.

The funding organisation (the Psoriasis Association) will support with recruitment by advertising the study on their website, on their various social media platforms, and in their monthly newsletter. Flyers will be displayed in Participant Identification Centers as well as on campus at King's College London. Social media will be used to promote the study and the study will also be advertised in the biweekly recruitment newsletter that is circulated to the staff and student population at King's College London.

Individuals responding to the study advertisements will be emailed an information sheet to evaluate if the METRED-P study is suitable for them. An eligibility video call will be arranged with the Research Nutritionist, to verify the volunteer meets the inclusion criteria, explain the information sheet and the informed consent process, and address any questions. Eligible respondents will be invited to an online video screening consultation on Microsoft Teams with the Research Nutritionist and Consultant Dermatologist to confirm their eligibility. The eligibility call and screening consultation will not be recorded and will be conducted confidentially, in a private office. Volunteers who meet the inclusion criteria will be invited to attend a screening clinic visit in the Metabolic Research Unit, 4th floor (Corridor A) at King's College London, 150 Stamford Street, SE1 9NH. The volunteer will be asked to complete the consent form and provide a fasted blood sample for a total of 13mL of blood (approximately 3.5 teaspoons) . A brief physical examination will be undertaken inclusive of weight, height, waist and hip circumference, body composition (% body fat) and clinic blood pressure. Participants will enrol in the the METRED-P study according to the inclusion and exclusion criteria and upon completing a 4-day diet diary assessment of habitual nutrient intake.

Eligible participants who passed the screening stages, will complete a hand-written 4-day diet diary and submit it by email to the Research Nutritionist prior to the initial clinic visit. Participants will arrive to the clinic at approximately 08:00AM, after a 12-hour overnight fast. A fasting blood sample will be taken intravenously for a total of 18mL of blood (approximately 4.5 teaspoons). Psoriasis severity will be assessed by the Consultant Dermatologist. Body composition and clinic blood pressure measures will be taken by the Research Nutritionist. Based on the pre-clinic 4-day diet diary, participants will receive personalised dietary guidance on their allocated dietary intervention, which should be adhered to for the duration of the study. On week 4 and week 8 of the study, virtual dietary consultation booster sessions will be arranged with the Research Nutritionist to reinforce the dietary advice and to maximise adherence with the allocated dietary interventions. Participants will also complete short multiple-choice questionnaires on the severity of their psoriasis. Wellbeing check-in calls are scheduled on week 2, week 6 and week 10 with the Research Nutritionist to ensure participant well-being and address any compliance issues. Participants will return for a clinic visit at the end of the study, to repeat the measures obtained at the initial visit and complete an exit questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* adults (aged 18 years or older)
* a medical diagnosis of plaque psoriasis
* a baseline Psoriasis Area Severity Index score between 5-10 (evaluated during screening)
* a Body Mass Index between 20-40
* not on tablet or injection therapies for psoriasis, OR if on tablet or injection therapies, is 6 months stable on the same dose of tablet or injection therapies

Exclusion Criteria:

* is taking Cyclosporine or Stelara in the past 3 months
* is receiving or has received photo (light) therapies for psoriasis in the past 3 months
* is a shift worker or is involved in shift work
* is planning on international travel during the study period
* is not weight stable or has attempted to lose weight during the past 6 months
* diagnosis of a gluten, nut, peanut, fish, or shellfish allergy
* diagnosis of a gluten or dairy intolerance
* is following a restrictive diet/restricting food groups i.e vegan, vegetarian, gluten-free , or a Mediterranean style diet
* is following any intermittent fasting regimes inclusive of 5:2, alternate day fasting or modified alternate day fasting, time-restricted eating over the past 6 months
* reports a habitual eating window < 12 h per day
* reports a baseline healthy diet (e.g. > 5 servings of fruits and vegetables per day, 1 serving of nuts per day , 2 servings of whole grains per day, 2 servings of fish per week, > 1 servings of nuts per day and rarely eats sweet snacks, cakes, fried foods and red meat).
* taking fish oil or other dietary supplements (except daily multivitamins providing no more than 200% of UK dietary recommended values)
* currently pregnant, currently breastfeeding or planning to become pregnant in the next 4 months
* is or has been diagnosed in the past with any of the following:

  * Anaemia
  * Asthma
  * Cancer in the last five years (except non-melanoma skin cancer)
  * Cardiovascular disease (angina, congenital heart disease, coronary artery disease, heat attack, heart failure or stoke)
  * Chronic gastrointestinal disease (Crohn's disease, ulcerative colitis, celiac disease or malabsorption diseases)
  * Chronic kidney disease
  * Dementia
  * Eating disorders (anorexia, bulimia or binge eating disorder)
  * Insulin dependent diabetes
  * Liver disease
  * Lupus
  * Multiple sclerosis
  * Rheumatoid arthritis
  * Thyroid disease
* history of bariatric surgery
* history of substance abuse or alcoholism (past history of alcohol intake >60 units/men or 50 units/women), within the last 12 months
* taking medication likely to interfere with study outcomes e.g. steroids (except occasional use of inhalers), anti-inflammatories or immune-suppressive drugs
* taking blood pressure medication, but has not been on a stable dosage during the last 3 months
* not on a stable topical treatment regimen for psoriasis (if prescribed)
* currently participating in a pharmaceutical study for psoriasis treatments (topical, light, tablet, or injection therapies) or has participated in a pharmaceutical study < 3 months ago
* currently participating in another diet intervention study or has participated in a diet intervention study < 3 months ago
* unwilling to record dietary intakes using handwritten diet diaries
* not fluent in the English language
* reports to have fainted in the past during an intravenous blood test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Average adherence to the diet intervention after 1 week, as assessed by the MEditerranean Diet Adherence Screener (MEDAS). | 1 week
  0-5 points = low adherence, 6-9 points = moderate adherence and 10-14 points = high adherence.
Average adherence to the diet intervention after 6 weeks, as assessed by the MEditerranean Diet Adherence Screener (MEDAS). | 6 weeks
  0-5 points = low adherence, 6-9 points = moderate adherence and 10-14 points = high adherence.
Average adherence to the diet intervention after 12 weeks, as assessed by the MEditerranean Diet Adherence Screener (MEDAS). | 12 weeks
  0-5 points = low adherence, 6-9 points = moderate adherence and 10-14 points = high adherence.

SECONDARY OUTCOMES:
The acceptability of the allocated dietary intervention, as assessed by participant records. | 12 weeks
  Expressed as rates of participant recruitment, attrition, and compliance.
The practicality of delivering the dietary interventions, as assessed with a exit questionnaire. | 12 weeks
  Expressed as the percentages of participant responses.

OTHER OUTCOMES:
Change between baseline and week 12 psoriasis severity, as assessed by the Psoriasis Area Severity Index (PASI). | 12 weeks
  0-4 = mild psoriasis, 5-10 = moderate psoriasis, and >10 = severe psoriasis.
Change in baseline self-reported psoriasis severity at 4 weeks, as assessed by the self-assessed Simplified Psoriasis Index (sa-SPI). | 4 weeks
  0-9 = mild psoriasis, 10-19 = moderate psoriasis and >20 = severe psoriasis.
Change in baseline self-reported psoriasis severity at 8 weeks, as assessed by the self-assessed Simplified Psoriasis Index (sa-SPI). | 8 weeks
  0-9 = mild psoriasis, 10-19 = moderate psoriasis and >20 = severe psoriasis.
Change in baseline self-reported psoriasis severity at 12 weeks, as assessed by the self-assessed Simplified Psoriasis Index (sa-SPI). | 12 weeks
  0-9 = mild psoriasis, 10-19 = moderate psoriasis and >20 = severe psoriasis.
Change between baseline and week 12 psoriasis severity, as assessed by the Physician's Global Assessment (PGA). | 12 weeks
  0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe.
Change in baseline self-reported psoriasis severity at 4 weeks, as assessed by the Dermatology Life Quality Index (DLQI). | 4 weeks
  0-1 points = no effect at all , 2-5 points = small effect , 6-10 points = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on the participant's life.
Change in baseline self-reported psoriasis severity at 8 weeks, as assessed by the Dermatology Life Quality Index (DLQI). | 8 weeks
  0-1 points = no effect at all , 2-5 points = small effect , 6-10 points = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on the participant's life.
Change in baseline self-reported psoriasis severity at 12 weeks, as assessed by the Dermatology Life Quality Index (DLQI). | 12 weeks
  0-1 points = no effect at all , 2-5 points = small effect , 6-10 points = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on the participant's life.
Change in baseline well-being at 4 weeks, as assessed by the World Health Organisation-5 (WHO-5). | 4 weeks
  0 represents the worst possible, and 25 representing best possible quality of life.
Change in baseline well-being at 8 weeks, as assessed by the World Health Organisation-5 (WHO-5). | 8 weeks
  0 represents the worst possible, and 25 representing best possible quality of life.
Change in baseline well-being at 12 weeks, as assessed by the World Health Organisation-5 (WHO-5). | 12 weeks
  0 represents the worst possible, and 25 representing best possible quality of life.
Change in baseline body weight, at 4 weeks, as assessed by self-measurement. | 4 weeks
  Calculated as the change between baseline body weight and body weight at week 4.
Change in baseline body weight at 8 weeks, as assessed by self-measurement. | 8 weeks
  Calculated as the change between baseline body weight and body weight at week 8.
Change in baseline body weight at 12 weeks, as assessed in clinic. | 12 weeks
  Calculated as the change between baseline body weight and body weight at 12 weeks.
Change in baseline Body Mass Index (BMI), as assessed by self-measurement. | 4 weeks
  Calculated as the change between baseline BMI and BMI at 4 weeks.
Change in baseline Body Mass Index (BMI), as assessed by self-measurement. | 8 weeks
  Calculated as the change between baseline BMI and BMI at 8 weeks.
Change in baseline Body Mass Index (BMI), as assessed in clinic. | 12 weeks
  Calculated as the change between baseline BMI and BMI at 12 weeks.
Change in waist-to-hip ratio. | 12 weeks
  Change between baseline and week 12 waist-to-hip ratio.
Change % body fat, as assessed by bioelectrical impedance analysis. | 12 weeks
  Change between baseline and week 12 body fat (%).
Change in % lean body mass, as assessed by bioelectrical impedance analysis. | 12 weeks
  Change between baseline and week lean body mass (%).
Change in clinic blood pressure. | 12 weeks
  Change between baseline and week 12 clinic blood pressure.
Change in fasting plasma glucose. | 12 weeks
  Change between baseline and week 12 fasting plasma glucose.
Change in fasting serum insulin. | 12 weeks
  Change between baseline and week 12 fasting serum insulin.
Change in fasting serum total cholesterol. | 12 weeks
  Change between baseline and week 12 fasting serum total cholesterol.
Change in fasting serum low density lipoprotein (LDL) cholesterol. | 12 weeks
  Change between baseline and week 12 fasting serum low density lipoprotein (LDL) cholesterol.
Change in fasting serum high density lipoprotein (HDL) cholesterol. | 12 weeks
  Change between baseline and week 12 fasting serum high density lipoprotein (HDL) cholesterol.
Change in fasting serum triglycerides. | 12 weeks
  Change between baseline and week 12 fasting serum triglycerides.
Change in fasting serum high-sensitivity C-Reactive Protein. | 12 weeks
  Change between baseline and week 12 fasting serum high-sensitivity C-reactive protein.
Change in fasting serum Tumour Necrosis Factor - alpha (TNF - α). | 12 weeks
  Change between baseline and week 12 fasting serum TNF - α.
Change in fasting serum Interferon - gamma (IFN - γ). | 12 weeks
  Change between baseline and week 12 fasting serum IFN - γ.
Change in fasting serum Interleukin - 6 (IL-6). | 12 weeks
  Change between baseline and week 12 fasting serum IL-6.
Change in fasting serum Interleukin - 12 (IL-12). | 12 weeks
  Change between baseline and week 12 fasting serum IL-12.
Change in fasting serum Interleukin - 17 (IL-17). | 12 weeks
  Change between baseline and week 12 fasting serum IL-17.
Change in fasting serum Interleukin - 17 (IL-23). | 12 weeks
  Change between baseline and week 12 fasting serum IL-23.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Hall, PhD, Principal Investigator — Reader in Nutritional Sciences
Locations (1):
- Metabolic Research Unit, Franklin-Wilkins Building, King's College London. 150 Stamford Street, Waterloo, London., London, Westminser, United Kingdom

REFERENCES:
- [Background] Ashcroft DM, Wan Po AL, Williams HC, Griffiths CE. Clinical measures of disease severity and outcome in psoriasis: a critical appraisal of their quality. Br J Dermatol. 1999 Aug;141(2):185-91. doi: 10.1046/j.1365-2133.1999.02963.x. PMID 10468786
- [Background] Pascoe VL, Enamandram M, Corey KC, Cheng CE, Javorsky EJ, Sung SM, Donahue KR, Kimball AB. Using the Physician Global Assessment in a clinical setting to measure and track patient outcomes. JAMA Dermatol. 2015 Apr;151(4):375-81. doi: 10.1001/jamadermatol.2014.3513. PMID 25549367
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Chularojanamontri L, Griffiths CE, Chalmers RJ. The Simplified Psoriasis Index (SPI): a practical tool for assessing psoriasis. J Invest Dermatol. 2013 Aug;133(8):1956-62. doi: 10.1038/jid.2013.138. Epub 2013 Mar 20. PMID 23807685